CLINICAL TRIAL: NCT06143280
Title: Functional Soft Palate Reconstruction
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-01689; mu23Schaefer2
Record Dates: First submitted 2023-11-08; First posted 2023-11-22 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Soft Palate Reconstruction
Keywords: swallowing phase; digastric muscle; palatal reconstruction; free radial flap plasty; displacement of the digastric muscle
MeSH Terms: interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Data collection — Data collection using entries in the medical records of the respective patients (surgery reports, progress notes, consultation reports, imaging and pathology reports) who underwent surgery with the new dynamic technique for soft palate reconstruction.

SUMMARY:
The aim of the study is to show that the innovative, dynamic palatal reconstruction technique (free radial flap plasty in combination with displacement of the digastric muscle) leads to a good functional outcome in terms of speech and swallowing in the context of the current literature.

DETAILED DESCRIPTION:
Tumors in the throat and pharynx are common and often lead to impaired swallowing and phonation after surgical tumor resection. The posterior part of the digastric muscle is responsible for sealing during the pharyngeal swallowing phase, among other things. By relocating the digastric muscle, a defect in the area of the soft palate can now be reconstructed with a muscle whose physiological function is already integrated into the complex process of the swallowing act and thus leads to a better seal. This new, previously undescribed reconstruction option has been used on various patients at the University Hospital with good functional results.

This study is to describe the new dynamic technique for soft palate reconstruction and to analyze the associated functional and surgical outcomes including postoperative complications, speech and swallowing function. The resulting values will be compared with the existing literature. The aim is to investigate whether the functional outcome in terms of phonation and swallowing can be improved by this technique.

ELIGIBILITY:
Inclusion Criteria:

* Patients after tumor resection of the soft palate with reconstruction by a free radial flap and displacement of the digastric muscle.

Exclusion Criteria:

* Patients with resected oropharyngeal carcinoma but without reconstruction using the dynamic technique described are excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Retrospective study of all patients who have undergone reconstruction of the soft palate with free radial flap plasty in combination with displacement of the digastric muscle between 2007 and 2017 at the University Hospital Basel.
Sampling Method: Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2023-11-06 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Number of complications | one time assessment at baseline
  Number of complications after reconstruction of the soft palate with free radial flap plasty in combination with displacement of the digastric muscle
Number of risk factors | one time assessment at baseline
  Number of risk factors in patients with reconstruction of the soft palate
Number of perioperative therapies (chemotherapy and radiotherapy) | one time assessment at baseline
  Perioperative therapies (chemotherapy and radiotherapy) in patients with reconstruction of the soft palate (descriptive)
Rate of different surgical indications | one time assessment at baseline
  Surgical indication in patients with reconstruction of the soft palate (descriptive)
Oncological status according to tumor, node, metastasis (TNM) classification | one time assessment at baseline
  Oncological status in patients with reconstruction of the soft palate (descriptive); TNM classification system for carcinoma is to establish the anatomic extent of the disease (Stage 0 - Indicates carcinoma in situ. Tis, N0, M0. Stage I - Localized cancer. T1-T2, N0, M0.
  Stage II - Locally advanced cancer, early stages. T2-T4, N0, M0. Stage III - Locally advanced cancer, late stages. T1-T4, N1-N3, M0.; Stage IV - Metastatic cancer. T1-T4, N1-N3, M1.)

CONTACTS AND LOCATIONS:
Overall Officials: Dirk J. Schaefer, Prof. Dr. med., Principal Investigator — Department of Plastic, Reconstructive, Aesthetic and Hand Surgery, University Hospital Basel
Locations (1):
- Department of Plastic, Reconstructive, Aesthetic and Hand Surgery, University Hospital Basel, Basel, Switzerland